CLINICAL TRIAL: NCT05723887
Title: The Effect of Attachment-Based Intervention Program on Attachment, Prenatal
Brief Title: Attachment-Based, Attachment, Prenatal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Collaborators: Tuba Uçar (Unknown)
Responsible Party: Principal Investigator, Esra SABANCI BARANSEL, Assistant professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020/605
Record Dates: First submitted 2023-01-13; First posted 2023-02-13 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Attachment Disorder
Keywords: prenatal distress; pregnancy; Midw,ifery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (ABIP group) (Experimental): The ABIP was created by the researchers in line with the literature and consisted of interventions that affect and increase prenatal attachment Gölbaşı et al., 2015; Güney & including perceiving /counting fetal movements, music therapy, preparation for the baby, writing notes/letters to the baby, watching images of the fetus/pregnancy. The program was completed in a total of five days, with one intervention per day. An ABIP kit, which contained the materials to be used by pregnant women during ABIP interventions, was provided to them by the researchers at the first meeting. ABIP intervention materials were included in the ABIP kit, using five different colored envelopes (Appendix 1). Pregnant women were also informed about the interventions and materials of ABIP by the researchers at the first meeting.
  Interventions: Behavioral: Attachment-Based Intervention Program
- control groups (No Intervention): No Intervention: Control group standard care group

INTERVENTIONS:
Behavioral: Attachment-Based Intervention Program — Attachment-Based Intervention Program
  Arms: Experimental (ABIP group)

SUMMARY:
This randomized controlled study was conducted in the pregnant outpatient clinics of a public hospital in Turkey. The sample of the study consisted of a total of 154 pregnant women (77 experiments, 77 controls). An attachment-based intervention program (ABIP) was applied to pregnant women in the experimental group. The ABIP included five interventions; (1) Perceiving/counting fetal movements, (2) Music therapy, (3) Preparation for the baby, (4) Writing notes/letters to the baby, and (5) Watching images of the fetus/pregnancy.

DETAILED DESCRIPTION:
This study aimed to determine the effect of attachment-based intervention program on attachment, prenatal expectation and stress level in pregnant women. This randomized controlled study was conducted in the pregnant outpatient clinics of a public hospital in Turkey. The sample of the study consisted of a total of 154 pregnant women (77 experiments, 77 controls). An attachment-based intervention program (ABIP) was applied to pregnant women in the experimental group. The ABIP included five interventions; (1) Perceiving/counting fetal movements, (2) Music therapy, (3) Preparation for the baby, (4) Writing notes/letters to the baby, and (5) Watching images of the fetus/pregnancy. The program was completed in a total of 5 days, one session per day.

ELIGIBILITY:
Inclusion Criteria:Communicating,

* Over the age of 18, and maimum age 40
* Pregnancy week between 24-40 weeks

Exclusion Criteria:

* Pregnant women with psychological diagnosis according to records

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 154 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Maternal Antenatal Attachment | one week
  It has a total of 19 items, focusing on pregnant women's feelings, attitudes and behaviors towards the fetus. This is a 5-point Likert type scale, scoring between 1 (the absence of feelings toward the fetus) and 5 (strong emotions toward the fetus).

SECONDARY OUTCOMES:
Prenatal Maternal Expectations | one week
  This is a 5-point Likert type scale, scoring from 1 (strongly agree) to 5 (strongly disagree). It consists of 34 items and two subscales: (1) Unrealistic Positive Prenatal Expectations (21 items measuring the mother's positive expectations about childbirth and motherhood role), (2) Unrealistic Negative Prenatal Expectations (13 items measuring the mother's negative expectations about childbirth and motherhood role).

OTHER OUTCOMES:
Revised Prenatal Distress Questionnaire | one week
  This is a three-point Likert-type scale, scoring from 0 (never) to 2 (very often). Total scale score ranges between 0 and 34. A higher total score indicates greater prenatal distress perceived by pregnant women.

CONTACTS AND LOCATIONS:
Overall Officials: Esra sabancı Baransel, asst. prof., Principal Investigator — esraa.sabancii@gmail.com
Locations (1):
- Esra Sabanci Baransel, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
individual participant data were not shared

REFERENCES:
- [Result] Golbasi Z, Ucar T, Tugut N. Validity and reliability of the Turkish version of the Maternal Antenatal Attachment Scale. Jpn J Nurs Sci. 2015 Apr;12(2):154-61. doi: 10.1111/jjns.12052. Epub 2014 Jun 24. PMID 24962076
- [Result] Pisoni C, Garofoli F, Tzialla C, Orcesi S, Spinillo A, Politi P, Balottin U, Tinelli C, Stronati M. Complexity of parental prenatal attachment during pregnancy at risk for preterm delivery. J Matern Fetal Neonatal Med. 2016 Mar;29(5):771-6. doi: 10.3109/14767058.2015.1017813. Epub 2015 Mar 9. PMID 25747945
- [Result] Yuksel F, Akin S, Durna Z. Prenatal distress in Turkish pregnant women and factors associated with maternal prenatal distress. J Clin Nurs. 2014 Jan;23(1-2):54-64. doi: 10.1111/j.1365-2702.2012.04283.x. Epub 2013 Jan 11. PMID 23305376